CLINICAL TRIAL: NCT05955339
Title: Comparing Healthcare Visit Recording and Open Notes to Improve the Chronic Illness Care Experience for Older Adults (The CHRONICLE Trial)
Brief Title: Comparing Healthcare Visit Recording and Open Notes to Improve Chronic iLlness Care Experience in Older Adults
Acronym: CHRONICLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other); Vanderbilt University Medical Center (Other); Beth Israel Deaconess Medical Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002056
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Audio Recording; Diabetes Mellitus; Hypertension; Patient-centered communication; Self-management; Older adults; Chronic conditions; After visit summary; Quality of life; Multimorbidity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to NOTES or NOTES+AUDIO using a block randomization technique with the clinician acting as the blocking variable. This strategy will ensure an equal number of patients per clinician will be randomly assigned to each study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOTES (Active Comparator): Patients in this arm will receive only the NOTES intervention.
  Interventions: Other: NOTES
- NOTES + AUDIO (Active Comparator): Patients in this arm will receive both the NOTES and AUDIO intervention.
  Interventions: Other: NOTES; Other: AUDIO

INTERVENTIONS:
Other: NOTES — The intervention will include: (1) a brief training on using the patient portal to access written visit information with assistance in setting up patient portal accounts where necessary (including strategies to share notes with a caregiver), (2) post-visit reminders to use the patient portal to access written visit information.
Other: AUDIO — The intervention will include: (1) audio recording all visits with the study clinician for six months, (2) training on how to record visits and access visit recordings, and (3) post-visit reminders listen to the visit recordings.
  Arms: NOTES + AUDIO

SUMMARY:
CHRONICLE is a randomized trial assessing the comparative effectiveness of providing written visit information via the patient portal (NOTES) versus NOTES plus visit audio recording (AUDIO) to older adult patients with chronic diseases on quality of life and other outcomes. During the trial, the team will also invite caregivers identified by patients to join the project.

DETAILED DESCRIPTION:
The research team is working with primary care clinics at three health systems across the country to enroll adults ages 65 and older who are managing diabetes or high blood pressure, plus one other disease. The team is assigning patients by chance to one of two groups. Each group will have an equal numbers of patients. Patients in one group will get access to visit notes through the patient portal. The research team will give patients guidance on how to find and use their visit notes. Patients in the other group will not only have access to their visit notes patients but also get access to audio-recordings of their visits. After each visit, patients in both groups will receive emails to review their visit information: 1) two days after their visit to remind them of their visit discussion and any tasks they may have, and 2) three days before their next visit, they will be asked to think of any changes from their last visit and to make a list of three things they want to talk to their doctor about. The team is comparing changes reported by patients over six months in quality of life, satisfaction, self-management ability, treatment adherence, and visit communication. The team will also invite caregivers identified by patients to join the project. They will show patients how to share their visit notes or recordings with caregivers. Caregivers will report on changes in how prepared they feel to provide care, burden related to caregiving, and how much they felt part of the patient's visit conversation.

ELIGIBILITY:
PATIENTS:

Inclusion Criteria:

* ≥ 65 years;
* With multimorbidity (diabetes or hypertension plus one of the following: arthritis (osteoarthritis and rheumatoid arthritis), asthma, atrial fibrillation, Alzheimer's disease and related dementia (not severe), cancer, chronic obstructive pulmonary disease, depression, heart disease, heart failure, hyperlipidemia, osteoporosis, kidney disease and stroke. Patients with diabetes plus hypertension are eligible.
* Have had two or more clinic visits in the previous 12 months;
* Plan on receiving ongoing care at the clinic with the enrolled clinician for the subsequent 6 months;
* Do not have vision or hearing problems that cannot be corrected; and
* Have not recorded a clinic visit for personal use in the past 6 months

Exclusion Criteria:

* With no capacity to consent to the project;
* With schizophrenia and other psychotic disorders, current substance-use disorders, uncorrected hearing or visual impairment;
* Living in skilled nursing homes or hospice, because they engage less in self-management;
* With cognitive impairment as identified by a score of ≤3 on the six-item screener (SIS)
* Lacking internet access;
* Who do not speak English or Spanish;
* Who (i) do not have access to a personal email, (ii) do not have an email address shared with a family member or patient-identified caregiver, and/or (iii) are not interested in creating a personal email as this would prevent them from engaging with the intervention(s); and
* Who do not wish to create a patient portal account, if they do not already have one as this would prevent them from engaging with the intervention(s).

CAREGIVERS:

Inclusion criteria:

* Agree to their identified role as a caregiver;
* Speak English or Spanish;
* Have capacity to consent to research participation; and
* ≥ 18 years.

Exclusion criteria:

* No capacity to consent to the project;
* Living in skilled nursing homes or hospice;
* Lacking internet access; or
* Do not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Quality of Life - Mental functioning | 6 months from enrollment
  Quality of life using Global PROMIS (Patient-Reported Outcome Measurement Information System) is a 10-item patient reported measure with two domains: mental and physical health. Domain scores range from 4 to 20, with higher scores representing better health.
Quality of Life - Physical functioning | 6 months from enrollment
  Quality of life using Global PROMIS (Patient-Reported Outcome Measurement Information System) is a 10-item patient reported measure with two domains: mental and physical health. Domain scores range from 4 to 20, with higher scores representing better health.

SECONDARY OUTCOMES:
Self-management ability | 6 months from enrollment
  Self-management ability using the Patient Activation Measure-Short Form is a 13-item patient reported measure. Scores are range from 0 (low activation) to 100 (high activation).
Medication adherence | 6 months from enrollment
  Medication adherence using Adherence to Refills and Medications (ARMS-7), an seven-item measure with two domains: i) medication taking and ii) medication refilling. ARMS-7 scores range from 7 (high adherence) to 28 (low adherence).
General satisfaction | 6 months from enrollment
  General satisfaction using the two-item general satisfaction sub-scale from the Patient Satisfaction Questionnaire-18 (PSQ-18). The subscale is scored as a mean of the two questions with a potential score ranging from 1 to 5. Higher scores indicate more satisfaction.
Visit communication style and shared decision-making | 6 months from enrollment
  Visit communication style and shared decision making using 14 items (6 of 7 subscales) from the Interpersonal Process of Care (IPC) survey. Each of the 6 subscales has a potential score of 1 to 5. Direction of the score depends on the subscale.

OTHER OUTCOMES:
Caregiver preparedness [Caregiver outcome] | 6 months from enrollment
  Caregiver preparedness using the 9-item Preparedness for Caregiving Scale. Scores range from 0 to 4 with higher scores corresponding to caregivers feeling more prepared for caregiving.
Caregiver burden [Caregiver outcome] | 6 months from enrollment
  Caregiver burden using the 10-item Burden Scale for Family Caregivers-Short Form (BSFC-s). BSFC-s scores range from 0 to 30 with higher scores indicating greater caregiver burden.
Caregiver engagement in clinic visit [Caregiver outcome] | 6 months from enrollment
  Caregiver engagement in clinic visit using the 12-item CAregiver Perceptions About CommunIcaTion with Clinical Team members (CAPACITY). Potential scores range from 12 to 48 with higher score indicating perceptions of better quality communication and capacity-assessment from the care team.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Barr, PhD, Principal Investigator — Dartmouth College; Kerri L Cavanaugh, MD, Principal Investigator — Vanderbilit University Medical Center; Meredith C Masel, PhD, Principal Investigator — University Texas Medical Branch
Locations (3):
- United States (3):
  - Dartmouth Hitchcock Clinics Manchester, Manchester, New Hampshire
  - Vanderbit University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of this research, the research data from this project will be deposited with the Patient-Centered Outcomes Data Repository (PCODR), based at the Inter-university Consortium for Political and Social Research (ICPSR), University of Michigan to ensure that the research community has long-term access to the data. This will include all deidentified data from surveys and/or transcripts from recorded interviews or encounters. For those who consent, we will also put identifiable recordings into the repository.
Supporting Information: Study Protocol, ICF
Time Frame: At the completion of data analysis.
Access Criteria: All access will be coordinated through PCODR/ICPSR.
URL: https://www.icpsr.umich.edu/web/pages/pcodr/about.html

REFERENCES:
- See also: Information about the CHRONICLE Trial — https://www.openrecordings.org/projects-chronicle